CLINICAL TRIAL: NCT02109432
Title: Short-term Behavior Change With Pedal Desk Installation
Acronym: PD-ST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Continued development of technology
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Corby K. Martin, Principal Investigator, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PBRC 2013-051
Record Dates: First submitted 2014-03-12; First posted 2014-04-09 (Estimated); Results first posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Physical Activity in the Workplace
Keywords: Pedal Desk; Physical Activity; Workplace; Energy Expenditure
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pedal Desk (Other): Participants will complete three 2-week conditions in the following order:
  1. Self-directed Pedal Desk
  2. Facilitated Pedal Desk
  3. Facilitated Pedal Desk with Pedometer
  Interventions: Behavioral: Self-Directed Pedal Desk; Behavioral: Facilitated Pedal Desk; Behavioral: Facilitated Pedal Desk with Pedometer

INTERVENTIONS:
Behavioral: Self-Directed Pedal Desk — participants will have a pedal desk installed in their office and will have access to their daily recorded data but will not have any other form of feedback or goal-setting
Behavioral: Facilitated Pedal Desk — participants are provided with their daily recorded pedal desk data and additional daily behavioral support from an interventionist (e.g., feedback and goal-setting) to increase their use of the pedal desk by an individually negotiated and agreed upon amount
Behavioral: Facilitated Pedal Desk with Pedometer — participants will be provided with their daily recorded pedal desk and step count data and additional daily behavioral support from an interventionist (e.g., feedback and goal-setting) to increase their use of the pedal desk by an individually negotiated and agreed upon amount and increase their step count by 3,000 steps/day compared to baseline.

SUMMARY:
The purpose of this investigation is to evaluate participant use of a dedicated office pedal desk with and without behavioral support.

DETAILED DESCRIPTION:
For this pilot study the investigators will identify and recruit up to 20 full time Pennington Biomedical staff members employed in sedentary jobs (i.e., report mostly sitting during working hours). The sample size is limited by the number of pedal desks being built for this pilot study and the need for timely data generation. Although the investigators can stagger starts as needed, all participants must intend to be on campus for the subsequent 6 weeks after they start the intervention. Two cohorts of 10 participants will complete the three 2-week conditions in the following order: 1) SELF-DIRECTED use where participants have access to their daily recorded data but will not have any other form of feedback or goal-setting; 2) FACILITATED use where participants are provided with their daily recorded pedal desk data and additional daily behavioral support from an interventionist (e.g., feedback and goal-setting) to increase their use of the pedal desk by an individually negotiated and agreed upon amount; 3) FACILITATED use with PEDOMETER where participants will be provided with their daily recorded pedal desk and step count data and additional daily behavioral support from an interventionist (e.g., feedback and goal-setting) to increase their use of the pedal desk by an individually negotiated and agreed upon amount and increase their step count by 3,000 steps/day compared to baseline. Participants will be asked to pedal at a sustainable and self-selected pace while using the pedal desk.

ELIGIBILITY:
Inclusion Criteria:

* Be a full-time employee at Pennington Biomedical Research Center
* Be between 21 and 65 years of age
* Primarily sit while at work
* Work from a private office/cubicle

Exclusion Criteria:

* Weigh more than 250 pounds
* Have physical limitations that prevent performance of pedaling motions
* Plan to be away from work for the 6 weeks of the intervention
* Be pregnant
* Have a pace maker and/or metal joint replacement
* Plan to be away from work for the 6 weeks of the intervention

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corby K Martin, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Pedal Desk: Three 2-week pedal desk conditions (Self-directed, Facilitated and Facilitated Pedal Desk with Pedometer)
Period: Overall Study
Arm/Group | Pedal Desk
Started | 7
Completed | 6
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Pedal Desk: Participants will complete three 2-week pedal desk conditions in the following order:
  1. Self-directed Pedal Desk
  2. Facilitated Pedal Desk
  3. Facilitated Pedal Desk with Pedometer
Arm/Group | Pedal Desk
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Weight Change (kg)
Description: KG weight change from Baseline to 6 weeks
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Pedal Desk
Number analyzed (Participants) | 6
kg | -.98 (1.09)

ADVERSE EVENTS:
Time Frame: 6 weeks of study participation
Description: adverse event collection was completed at clinic visits. The standard clinical trials definition of AEs was used.
Arm/Group | Pedal Desk
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
The study's progress was hindered by technical problems with the pedaldesk's software that limited the ability of participants and staff members to view pedaldesk data. This hindered deployment of the anticipated 3 levels of support.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes